CLINICAL TRIAL: NCT03235934
Title: Glycemic Impact on Glioblastoma Outcomes
Status: Withdrawn | Type: Observational
Why Stopped: Logistical Issues
Sponsor: University Health Network, Toronto (Other)
Collaborators: Sinai Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 15-9329
Record Dates: First submitted 2017-07-18; First posted 2017-08-01 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Glioblastoma Multiforme; Hyperglycemia
Keywords: glucose monitoring
MeSH Terms: conditions — Glioblastoma; Hyperglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This pilot study aims to evaluate the feasibility of close glucose monitoring and management of patients (targeting fasting and pre-meal glucose of 4-7 mmol/L) using state-of-the-art flash glucose monitoring (FGM) technology. The glycemic intervention will be personalized based on individual blood glucose levels. Although the glycemic interventions used in this study include standard medications and methods of glucose monitoring used for patients with diabetes, this pilot study will specifically evaluate the feasibility of using these approaches in patients with GBM, appreciating their additional medical, functional and social challenges.

DETAILED DESCRIPTION:
The purpose of this pilot study is to determine the feasibility of using close monitoring and management of glucose levels in patients undergoing radiation and chemotherapy for glioblastoma.

The glucose management will include the use of standard metformin a common treatment for patients with early type 2 diabetes that has also shown anti-tumor effects in GBM, and will be further personalized based on individual blood glucose levels. Additional anti-hyperglycemic management will be provided at the discretion of the Endocrinologist.

Close glucose monitoring will include flash glucose monitoring (FGM) with a device called an FreeStyle Libre Pro Flash Glucose Monitoring System, finger-prick glucose measures (standard approach for patients with diabetes) and weekly blood tests (our current standard for patients with GBM).

In addition to determining the feasibility of using these approaches, this pilot study will help identify the simplest and most effective approach of managing glucose levels in patients with GBM appreciating their additional medical, functional and social challenges.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (> 18 years old) with a new histologically-confirmed diagnosis of glioblastoma who are planned to receive a 6-week course of concurrent radiation and temozolomide
* Has evidence of random glucose of at least 7.8 mmol/L or fasting blood glucose of at least 6.1 mmol/L (meeting criteria for oral diabetic medications)
* Able to provide informed consent
* Able to understand and follow instructions regarding self-administered capillary glucose measurements

Exclusion Criteria:

* Contraindication to MRI with gadolinium
* Taking anti-hyperglycemic medications at the time of study eligibility screen
* Unable to participate in neurocognitive evaluation in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who are newly diagnosed with glioblastoma
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2019-10-01 (Estimated); Study Completion 2020-01-24 (Actual)

PRIMARY OUTCOMES:
Total time spent in target glucose level | 1 week
  total time spent in target range of 4-10 mmol/L based on FGM data during week 6 of radiotherapy and temozolomide therapy

SECONDARY OUTCOMES:
Area under the curve for glycemic exposure and variability | baseline, week 1, 2, 3, 4, 5, 6, 10-13, 3 months
  Glucose levels measured using FGM vs conventional clinical measures (e.g. capillary blood glucose)
Neurocognitive Function | Baseline
  To explore the association between glycemia and neurocognitive functions patients will undergo standardized tests
Neurocognitive Function | After week 10 and before week 13
  To explore the association between glycemia and neurocognitive functions patients will undergo standardized tests
Neurocognitive Function | 3 month follow up visit
  To explore the association between glycemia and neurocognitive functions patients will undergo standardized tests
prevalence of sensor site problems | From baseline to week 6 - the time from sensor insertion through completion of study intervention
  infection, irritation, and secondary complication in the study cohort

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No